CLINICAL TRIAL: NCT03245788
Title: Pilot Project to Better Understand Non-Clinical Needs of Cancer Patients
Brief Title: Effectiveness of Lay Navigators in Meeting Cancer Patients' Non-Clinical Needs: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marcy Winget, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 42674
Record Dates: First submitted 2017-05-04; First posted 2017-08-10 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Gynecologic Cancer; Neck Cancer; Head and Neck Cancer; Gastrointestinal Cancer; Thoracic Cancer; Cutaneous Tumor; Urologic Cancer; Neurologic Cancer; Lymphoma; Sarcoma; Bone Marrow Transplant
Keywords: Lay Navigator; Quality of Care; High-Need Cancer Treatment Regimen
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Skin Neoplasms; Urologic Neoplasms; Lymphoma; Sarcoma

STUDY DESIGN:
Intervention Model Description: There will be 12 groups in each arm which reflects the 12 different cancer types.
Masking Description: No masking occurs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lay Navigation (Experimental): Patients with even MRN.
  Interventions: Other: Lay Navigation
- Usual Care (No Intervention): Patients with odd MRN.

INTERVENTIONS:
Other: Lay Navigation — Patients who are assigned to intervention will be contacted by a navigator who will explain and offer their services to the patient. Navigators focus efforts on supporting patients in self-management and in supporting non-medical needs.
  Arms: Lay Navigation

SUMMARY:
The Stanford Cancer Center is undertaking a Transformation Initiative in order to improve the quality of care and care coordination across the continuum of care. The newest innovation is to introduce lay navigators to specified high-need patients. The larger goal of the project is to assess whether lay navigators can address non-clinical patient needs in a timely fashion and appropriately connect them with their clinical team when warranted. It is expected that proactive interaction with patients will decrease patient anxiety/stress related to their cancer and facilitate higher patient engagement and improved management of physical, social,and emotional health. For the pilot project, the smaller goal is to understand: how lay navigator time is used; the types and frequency of issues brought up by patients; resources that patients are given or referred to; type and frequency of mode of contact with patients; and patients' acceptance of navigators based on refusal. An electronic intake form will be used to collect this information so that data can be analyzed regularly to inform changes to the navigator program as needed.

DETAILED DESCRIPTION:
The Stanford Cancer Institute is undergoing a 5-year Transformation Initiative that began in 2013. One of the goals of this initiative is to increase patient engagement. The underlying premise is that engaged patients will be more likely to attend all their visits, receive all their treatments, and understand ways to manage treatment side effects so that they are less likely to go to the emergency room (ER) or be admitted to the hospital. An approach being tested is to use lay navigators to help identify patient issues and help them address the issues through a combination of direct supportive activities (e.g., calling clinical team for the patient) and activities that help the patients help themselves (helping them understand when side effects warrant a call to their clinical team that they make themselves).

Information including patient acceptance/refusal of navigator services; number and types of contacts with patients (phone, in-person, email); types of issues discussed (financial, social, educational, physical, emotional, etc); referrals made; and time spent with patients for each encounter will be routinely entered by the navigators for each patient contact. The data entered will be evaluated regularly to closely monitor navigator activities and better understand cancer patient issues/needs. This information will be used to inform possible training needs of navigators, educational needs of patients,needs for better referral support,help predict navigator case-load, and other issues.

Eligibility Criteria:

All new biopsy positive cancer patients that have a treatment plan to receive at least 2 treatment modalities: surgery, chemotherapy and/or radiation therapy at Stanford are eligible. Because there will be more patients eligible than the navigators can manage, only patients with an even MRN will receive a navigator for the pilot. The overall purpose of the pilot is to learn which patients benefit most and which services navigators are able to best help with. The investigators expect the pilot to last 6-12 months. Mixed methods will be used to evaluate the navigators and will include existing patient experience surveys, unscheduled hospitalizations, ER visits, interviews with patients, staff (including navigators), and physicians regarding their experience with and perceived value of navigators.

ELIGIBILITY:
Inclusion Criteria:

* New patient to eligible Cancer Care Program (CCP)
* Biopsy positive
* Plan to receive at least one treatment modality at Stanford: surgery, chemotherapy and/or radiation therapy
* Cancer that is treated by any of the following CCPs: Breast, Gynecologic oncology, Head/neck, Cutaneous (melanoma only), Thoracic, Gastrointestinal
* Patient has even numbered MRN

Exclusion Criteria:

* Anyone with odd numbered MRN
* Anyone in other cancer programs that are not included
* Biopsy negative
* No treatment modality received
* Patients with already established care/treatment i.e. not new patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Experience/Satisfaction: Difference in topbox scores | 3-18 months after eligibility is determined
  Difference in topbox scores from apriori selected questions from the transformation evaluation in navigated vs not navigated patients.
Rates of unplanned hospitalization and ER visits | 0-18 months after eligibility is determined
  Comparison of rates of unplanned hospitalizations and ER visits among eligible patients in the navigated group vs. un-navigated patients.

SECONDARY OUTCOMES:
Utilization of non-treatment-related cancer services | 0-18 months after eligibility is determined
  Comparison of the proportion of navigated patients that used non-treatment-related cancer services to those not navigated. Examples of services include palliative care, supportive care, nutrition, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Asch, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hennink MM, Kaiser BN, Marconi VC. Code Saturation Versus Meaning Saturation: How Many Interviews Are Enough? Qual Health Res. 2017 Mar;27(4):591-608. doi: 10.1177/1049732316665344. Epub 2016 Sep 26. PMID 27670770
- [Background] O'Cathain A, Murphy E, Nicholl J. Three techniques for integrating data in mixed methods studies. BMJ. 2010 Sep 17;341:c4587. doi: 10.1136/bmj.c4587. No abstract available. PMID 20851841
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Derived] Winget M, Holdsworth L, Wang S, Veruttipong D, Zionts D, Rosenthal EL, Asch SM. Effectiveness of a Lay Navigation Program in an Academic Cancer Center. JCO Oncol Pract. 2020 Jan;16(1):e75-e83. doi: 10.1200/JOP.19.00337. Epub 2019 Oct 24. PMID 31647691